CLINICAL TRIAL: NCT03890393
Title: Muscle Activity of Pericranial Muscles in Patients With Episodic or Chronic Headache vs Asymptomatic Controls: a Cross-sectional Study
Brief Title: A Clinical Observation on Electrophysiology in Headache Patients With Myofascial Trigger Points
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-SR-037
Record Dates: First submitted 2019-02-12; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Myofascial Trigger Points
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with episodic headache
  Interventions: Device: Electromyography
- patients with chronic headache
  Interventions: Device: Electromyography
- healthy controls
  Interventions: Device: Electromyography

INTERVENTIONS:
Device: Electromyography — Muscle activity was bilaterally tested with needle electromyography at rest status, targeting at myofascial trigger points (MTrPs) in the frontal, temporal, sternocleidomastoid (SCM), splenius capitis, splenius cervicis and trapezius of each subject.

SUMMARY:
Through an observational, cross-sectional study, muscle activity was compared among 21 subjects with episodic headache, 17 subjects with chronic headache and 17 age-matched healthy controls. Muscle activity was bilaterally tested with needle electromyography at rest status, targeting at myofascial trigger points (MTrPs) in the frontal, temporal, sternocleidomastoid (SCM), splenius capitis, splenius cervicis and trapezius of each subject. Headache characteristics (intensity, frequency and duration), McGill Pain Questionnaire (MPQ) and Digital Span (DS) scales were secondary outcomes. The correlation between muscle activity and headache characteristics was also analyzed.

This study provides preliminary evidence of the relationship between muscle and the chronicity of headache.

ELIGIBILITY:
Inclusion Criteria:

1. Have at least one onset of headache in the last week,
2. Aged between 18-65 years,
3. No special treatment or invasive test on pericranial muscles in the last month, and no painkillers or muscle relaxants in the last week.

Exclusion Criteria:

1. History of surgery, trauma, tumor and spinal disease affecting the head and neck,
2. Being unable to cooperate with inspection and questionnaires for any reason (severe systemic disease, bleeder, communication barriers and so on),
3. People with definite mental disorders such as anxiety and depression.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the patients were recruited from the headache clinic of Neurology in the first affiliated hospital of Nanjing Medical University from January/2018 to October/2018. Their diagnosis of headache were made according to the third edition of International Classification of Headache Disorders (ICHD-III).
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Pericranial muscle activity | On the day the participant was enrolled
  It was evaluated with EMG/EP equipment(9031A070 KEYPOINT Dantec) and the matching disposable needle electrode(Specification: 25mm*0.3mm, 30G) with a sampling frequency of 125 Hz and a measuring range of 0.2mv.The spontaneous electric activity of each pericranial muscle was recorded as 0 to 4 scores: 0 score= no repeatable spontaneous electric activity, 1 score=a single, repeatable string of spontaneous electric activity, 2 scores= obvious spontaneous electric activity in two or more areas of the muscle, 3 scores= obvious spontaneous electric activity in any area of the muscle, 4 scores= a lot of spontaneous electric activity over the whole record screen. The maximum scores of a participant was 48(6*2*4［insertion(frontal, temporal, sternocleidomastoid, splenius capitis, splenius cervicis and trapezius) *right or left* maximum scores of a muscle]).

SECONDARY OUTCOMES:
Short Form of the McGill Pain Questionnaire(SF-MPQ) | Immediately after the enrollment
  This scale included three parts:Pain Rating Index (PRI), a 10cm-visual analogue scale(VAS) and Present Pain Intensity (PPI).PRI included 15 items to describe the characteristics of the pain(like nature and emotional problems) and each item was assessed with 0-3 scores.The higher scores respresented more serious condition.Total points of PRI was 0-15*3.VAS relefected their average intensity of the headache during the last month and was recorded as 0-10 scores according to the length.The higher scores respresented more serious average pain;PPI was recorded as 0-5 scores and the higher scores respresented more serious present pain(0 point=no pain;1 point=a little uncomfortable;2 points=uncomfortable;3 points=obvious headache;4 points=serious headache;5 points=unbearable headache).Total scores of SF-MPQ= PRI +VAS +PPI.
Digital Span Test | Immediately after the enrollment
  Participants were requested to recite along and against two independent digits,seperately having 2-13 and 2-10 numbers.The highest number of the digits they recited was the score((2+2)-(13+10)) and the more scores they got, the wider memory they had.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Qi, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China